CLINICAL TRIAL: NCT05010278
Title: Evaluation of Factors Associated With Return to Sports Activity Six Months After Anterior Shoulder Stabilisation With Latarjet.
Acronym: ERASME
Status: Completed | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Other Study IDs: COS-RGDS-2020-06-024
Record Dates: First submitted 2021-08-16; First posted 2021-08-18 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Shoulder Luxation
MeSH Terms: conditions — Shoulder Dislocation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Latarjet: Patients followed up 6 months after a Latarjet procedure
  Interventions: Procedure: Latarjet

INTERVENTIONS:
Procedure: Latarjet — Patients followed up 6 months after a Latarjet procedure

SUMMARY:
On a population of sports patients who had undergone a Latarjet operation for post-traumatic anterior shoulder instability, reviewed in consultation 6 months after the operation as part of an ordinary follow-up and divided into two groups according to their current sports practice.

Group 1: "SUCCESS": return to the same level in the same sport. Group 2: "FAILURE": return to the same sport with a reduced level or change of sport or significant reduction or cessation of sporting activity.

DETAILED DESCRIPTION:
Primary objective:

to assess the impact of patients' psychological state on failure to return to sport.

Secondary objectives:

* To compare the functional assessment of the shoulder of patients for whom return to sport is successful or unsuccessful (Walch score, isokinetic tests and CKCUES Test score)
* To describe the factors associated with failure to return to sport

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older, having been informed of the research
* Sports patients who have expressed their desire to resume their sporting activity
* Patient who has undergone a first intention Latarjet operation
* Patient regularly monitored since the operation and for whom all the data collected during the six-month follow-up visit are available

Exclusion Criteria:

* Patient operated for revision surgery
* Patient with an associated rotator cuff or biceps injury
* Patient under court protection, guardianship or curatorship
* Patient who has indicated his opposition to the use of his medical data (by completing and returning the non-opposition form which will be sent to him)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed up 6 months after a Latarjet procedure.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
SISRI score | 6 months
  The Shoulder Instability-Return to Sport after Injury (SIRSI) score will be compared between groups by a Student's t test or by a non-parametric Mann-Whitney test.

SECONDARY OUTCOMES:
Walch-Duplay Score for Instability of the Shoulder | 6 months
  Walch-Duplay Score for Instability of the Shoulder
Isokinetic test: peak force | 6 months
  peak force (in newton-metre)
Isokinetic test: relative peak force | 6 months
  relative peak force: peak force/body weight (in newton/kilogram)
Isokinetic test: eccentric peak force | 6 months
  eccentric peak force achieved in external stroke
Closed kinetic chain upper extremity stability (CKCUES) test | 6 months
  The Closed Kinetic Chain Upper Extremity Stability Test (CKCUEST) is a tool developed and used in the clinic to evaluate progress during upper extremity rehabilitation. A need exists for reference values of CKCUEST for use in a clinical setting.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre HARDY, MD, Principal Investigator — Clinique du sport
Locations (1):
- Clinique du Sport, Paris, France

IPD SHARING:
Plan to Share IPD: No